CLINICAL TRIAL: NCT01628939
Title: Association Between Clinical Signs Assessed by Manual Segmental Examination and Findings of the Lumbar Facet Joints in Magnetic-resonance Scans in Subjects With and Without Current Low Back - a Prospective Single-blinded Study
Brief Title: Association Between Clinical Signs and MRI Findings of the Lumbar Facet Joints
Status: Completed | Type: Observational
Sponsor: Christoph Maier, Prof. Dr. (Other)
Responsible Party: Sponsor-Investigator, Christoph Maier, Prof. Dr., Prof. Dr. med., Head of the Department of Pain medicine, Ruhr University of Bochum
Organization: Ruhr University of Bochum (Other)
Other Study IDs: FacetJointEdema2009
Record Dates: First submitted 2012-06-17; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Low Back Pain; Facet Joint Pain
Keywords: low back pain; facet joint pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- current low back pain: subjects with current low back pain (i.e. more than 30 days of low back pain in the last three months)
  Interventions: Other: MRI of the lumbar spine; Other: manual segmental examination of the lumbar facet joints
- controls: subjects with less than 30 days of low back pain in the last three months
  Interventions: Other: MRI of the lumbar spine; Other: manual segmental examination of the lumbar facet joints

INTERVENTIONS:
Other: MRI of the lumbar spine — standard protocol, approximately 30 minutes
Other: manual segmental examination of the lumbar facet joints — use of three different segmental facet joint provocation tests (spinal palpation, segmental rotation and springing-test) from Th12-L1 to L5-S1

SUMMARY:
The purpose of this study is to determine

1. the prevalence of lumbar facet joint pain detected by manual segmental provocation tests
2. the prevalence of MRI findings of the lumbar facet joints (hypertrophy, effusion, edema)
3. the association of lumbar facet joint pain and MRI findings on a segmental level

in subjects with current low back pain and in a control group.

ELIGIBILITY:
Inclusion Criteria for both study groups:

* age > 18
* written informed consent
* ability to perform required examinations

Inclusion Criterion for current low back pain-group:

- more than (>=) 30 days of low back pain in the last three months

Inclusion Criterion for control group:

- less than 30 days of low back pain in the last three months

Exclusion Criteria for both study groups:

* acute radicular low back pain in the last three months
* claustrophobia
* spondylodesis of the lumbar spine
* any metallic implants which are not MRI-compatible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pain clinic, sports clubs and fitness centers
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Number of facet joints per person which show facet joint pain and FJ effusion and/ or edema | 2 hours
  association of facet joint pain and MRI facet joint findings is determined

SECONDARY OUTCOMES:
number of painful facet joints per person | 2 hours
  prevalence of facet joint pain assessed by manual segmental provocation tests
number of facet joints diagnosed with facet joint effusion and/ or edema per person | 2 hours
  prevalence of facet joint findings in the lumbar spine assessed by MRI (facet joint effusion and/ or facet joint edema)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, M.D., PhD, Study Director — Head of the Department of Pain medicine, BG Universitätsklinikum Bergmannsheil GmbH, 44789 Bochum, Germany
Locations (1):
- Department of Pain Medicine, BG Universitätsklinikum Bergmannsheil GmbH, Bochum, North Rhine-Westphalia, Germany